CLINICAL TRIAL: NCT04915196
Title: Investigation of Efficacy and Gastrointestinal Tolerability of Liposomally Bound Iron Compared to Ferrous Sulphate in Women With Abnormal Uterine Bleeding
Brief Title: Tolerability of Iron Therapy in Women With AUB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB20-1546
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Iron Deficiency Anemia; Abnormal Uterine Bleeding
MeSH Terms: conditions — Anemia, Iron-Deficiency; Metrorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ferrous Sulphate: Women age 18-50 yo that have been diagnosed with iron deficiency anemia secondary to abnormal uterine bleeding using Ferrous Sulphate for iron replacement
  Interventions: Dietary Supplement: Liposomally-bound Iron
- Liposomally-bound Iron: Women age 18-50 yo that have been diagnosed with iron deficiency anemia secondary to abnormal uterine bleeding using Liposomally-bound Iron for iron replacement
  Interventions: Dietary Supplement: Liposomally-bound Iron

INTERVENTIONS:
Dietary Supplement: Liposomally-bound Iron — Ferric pyrophosphate microencapsulated in liposomal form is an over the counter natural health product approved by Health Canada and commonly used for iron replacement. If this product is prescribed as part of usual management of iron deficiency and patients consent to participation they will be contacted by telephone survey of gastrointestinal tolerability.

SUMMARY:
Telephone surveys of female patients using liposomally-bound iron and traditional iron sulphate preparations for the management of iron deficiency anemia to determine gastrointestinal tolerability.

DETAILED DESCRIPTION:
1. Rationale and Background:

   Abnormal uterine bleeding (AUB) affects women worldwide. In high income countries, heavy menstrual bleeding (a subset of AUB) is the most common cause of iron deficiency (ID) and iron deficiency anemia (IDA). Although estimates vary, it appears that 20-30% of IDA is a result of heavy menstrual bleeding. Oral iron replacement is a common treatment modality among patients diagnosed with IDA. However, traditional oral iron preparations commonly result in significant gastrointestinal side effects due to the metabolism of the complex that the iron is bound to. Gastrointestinal side effects related to iron therapy, including: metallic taste, nausea, flatulence, constipation, diarrhea, epigastric distress, vomiting, and melena. Therefore, liposomally bound iron is thought to provide a better side effect profile due to avoiding these traditional complexes. In theory, this will lead to higher rates of compliance and treatment efficacy if patients are not experiencing these side effects. Although we have limited data on the efficacy of this iron preparation, the literature suggests that other types of liposomally bound medications have similar efficacy as traditional preparations. Therefore, we believe that liposomally bound iron will provide an effective and well tolerated option for women suffering from IDA secondary to AUB.
2. Research Question and Objectives:

   How does a novel liposomally-bound iron therapy compare to ferrous sulphate in women with anemia secondary to abnormal uterine bleeding? 2a. Determine if it has less gastrointestinal side effects than ferrous sulphate 2b. Determine if it has similar efficacy to ferrous sulphate in correcting anemia secondary to abnormal uterine bleeding
3. Methods:

Pre-menopausal women, diagnosed with anemia secondary to abnormal uterine bleeding Recruitment via physician offices of gynecologists in Calgary, AB Two treatment arms, n=10 per arm Ferrous sulphate compared to treatment arm (liposomally bound iron) Baseline hemoglobin prior to iron therapy initiation Pre-op hemoglobin to compare efficacy of iron therapy Phone interview with patients using standardized, validated questionnaire to collect information regarding gastrointestinal side effects

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with iron deficiency secondary to abnormal uterine bleeding

Exclusion Criteria:

* Postmenopausal, premenarchal and pregnant women are excluded, as they do not have regular uterine bleeding associated with menses.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Nongravid women age 18-50 yo that have been diagnosed with iron deficiency secondary to abnormal uterine bleeding
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Subjective tolerability of oral administration | 8 weeks
  Survey of gastrointestinal reactions to iron replacement

SECONDARY OUTCOMES:
Hemoglobin | 8 weeks
  Relative change of hemoglobin
Hematocrit | 8 weeks
  Relative change of hematocrit
Ferritin | 8 weeks
  Relative change of ferritin

CONTACTS AND LOCATIONS:
Overall Officials: Chandrew Rajakumar, M.D., Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Background] Pereira DI, Couto Irving SS, Lomer MC, Powell JJ. A rapid, simple questionnaire to assess gastrointestinal symptoms after oral ferrous sulphate supplementation. BMC Gastroenterol. 2014 Jun 4;14:103. doi: 10.1186/1471-230X-14-103. PMID 24899360